CLINICAL TRIAL: NCT05207748
Title: The Relationship of Bone Mineral Density With Balance, Functional Ambulation and Falls in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Assoc. Prof, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E1/1026/2020
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Stroke Patients
Keywords: stroke; osteoporosis
MeSH Terms: conditions — Stroke; Osteoporosis | interventions — Bone Density

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with a history of falls: Demographic characteristics and medical histories (age, height, weight, smoking, alcohol use, comorbidities, medications, stroke onset date, stroke side, total number of rehabilitation received, assistive device use, history of falls) of all patients participating in the study will be recorded.
  Detailed physical examinations (mini-mental status assessment, brunstrum stages, spasticity assessments, orthosis use) will be performed. Berg Balance Scale, which will reveal the balance states; Functional ambulation scores and Timed Up and Go test will be applied to determine their functional status. In addition, the International Fall Efficiency Scale questionnaire will be administered. Bone mineral density will be evaluated to assess patients' bone health.
  Interventions: Diagnostic Test: Bone mineral density
- patients without a history of falls: Demographic characteristics and medical histories (age, height, weight, smoking, alcohol use, comorbidities, medications, stroke onset date, stroke side, total number of rehabilitation received, assistive device use, history of falls) of all patients participating in the study will be recorded.
  Detailed physical examinations (mini-mental status assessment, brunstrum stages, spasticity assessments, orthosis use) will be performed. Berg Balance Scale, which will reveal the balance states; Functional ambulation scores and Timed Up and Go test will be applied to determine their functional status. In addition, the International Fall Efficiency Scale questionnaire will be administered. Bone mineral density will be evaluated to assess patients' bone health.
  Interventions: Diagnostic Test: Bone mineral density

INTERVENTIONS:
Diagnostic Test: Bone mineral density — Bone mineral density (BMD) will be measured on the lumbar spine (L1-L4) and femoral neck by dual X-ray absorptiometry (DXA) method.

SUMMARY:
The aim of this study is to investigate the relationship between bone mineral density and balance, functional ambulation and falls in hemiparetic patients with stroke in the subacute and chronic phases.

DETAILED DESCRIPTION:
Improving balance function is considered as an important method for reducing the risk of falling after stroke and protecting bone health. Bone mineral density, a measure of bone health, has been reported to decrease after stroke, consistent with increased bone resorption and decreased bone formation. The aim of this study is to investigate the relationship between bone mineral density and balance, functional ambulation and falls in hemiparetic patients with stroke in the subacute and chronic phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 50 and ≤ 75 years old
* Patients with a 10-year risk of hip fracture ≥3%, major osteoporotic fracture risk ≥20% according to the Fracture Risk Assessment Tool, FRAX, scoring
* Patients with unilateral hemiplegia as a result of first-time stroke (onset time > 3 months)
* Patients who can stand for at least 2 minutes independently/under supervision for measurements while standing, and who can walk at least 10 meters independently/under supervision with or without walking aid for measurements taken while walking
* Patients whose cognitive status is able to understand the study instructions (Mini-Mental State Assessment score ≥ 23)
* Patients with stable medical and psychological status
* Patients willing to participate in the study

Exclusion Criteria:

* Patients with serious cardiovascular or musculoskeletal problems that prevent walking
* Patients with severe vision, hearing and language problems
* Patients with other neurological (Parkinson's, epilepsy, meningitis, cerebellar disease, vertigo, dizziness, polyneuropathy, etc.) or musculoskeletal (severe low back pain, knee problems) diseases that may affect balance performance other than stroke.
* Patients with peripheral vascular disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 patients
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | baseline
  Bone mineral density (BMD) will be measured on the lumbar spine (L1-L4) and femoral neck by dual X-ray absorptiometry (DXA) method.

SECONDARY OUTCOMES:
Berg Balance Scale | baseline
  The Berg Balance Scale is a widely used clinical test that can reveal a person's static and dynamic balance abilities. Total test score range from 0 (lowest balance) to 56 (highest balance) ability.
Functional Ambulation Classification | baseline
  The Functional Ambulation Classification is a functional walking test that evaluates ambulation ability. It includes six different categories and assesses ambulation status by determining how much support the patient needs while walking, regardless of whether they use assistive devices.
Timed up and go test | baseline
  The timed up and go test is a test used to evaluate mobility, balance, and walking in people with balance disorders.
Falls Self-Efficacy Scale | baseline
  The International Fall Activity Scale is a scale that examines an individual's concerns about the possibility of falling during 16 different activities that do not threaten daily life.The response option ranged from 1-4 depicted by 1 for being not at all concerned, 2 for being somewhat concerned, 3 for being fairly concerned and 4 for being very concerned.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided